CLINICAL TRIAL: NCT06799728
Title: Uterus Transplantation: Acceptability of the Procedure in Eligible Patients
Status: Active, not recruiting | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Other Study IDs: ACCUTX-20
Record Dates: First submitted 2024-12-30; First posted 2025-01-29 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2024-11

CONDITIONS: Focus: Uterus Transplant Procedure; Acceptability of the Uterus Transplantation Procedure
Keywords: Transplantation of the uterus

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
This study aims to define the knowledge and acceptability of uterine transplantation in patients suffering from infertility due to congenital or acquired absence of this organ, which are followed up in the U.O.C. of Gynecology and Pathophysiology of Human Reproduction Polyclinic S. Orsola-Malpighi and registered with the Italian Association for Androgen Insensitivity and Similar Conditions-AISIA.

DETAILED DESCRIPTION:
Absolute infertility from uterine factor (AUFI) is the term used to indicate the condition of women who cannot achieve pregnancy due to congenital or acquired absence of the uterus or the presence of an anatomically or physiologically non-functional utery1.

The causes of AUFI can be classified in primary/congenital (Mayer-Rokitansky-Kuster-Hauser-MRKH syndrome, Complete insensitivity to androgens-CAIS) and secondary/acquired (Asherman syndrome, previous hysterectomy for benign/malignant gynecological pathologies).

This condition was considered without therapeutic options until a few years ago, when the first birth from living donor uterus transplant was obtained (Sweden, 2014)2.

There are many challenges to the transplantation of the uterus:

* Ethical, complex and evolving issues: first of all the acceptability by patients;3
* the definition of inclusion criteria for donors and recipients, based on the results of procedures carried out to date;4
* the presence of the donor: deceased or living, and in the latter the use of minimally invasive surgical techniques5.

Primary objective of the study Define the acceptability of the uterus transplant procedure in the target population through a cross-sectional observational study using a targeted questionnaire.

Secondary objective To assess the knowledge of certain aspects of uterine transplantation among the population affected by SVCD. To identify the opinion and needs of the study population.

Expected results The information will help improve the efficiency and quality of health services for people with SVD.

ELIGIBILITY:
Inclusion Criteria:

* - age 18-44 years
* patients with AUFI (MRKH, CAIS, previous hysterectomy due to benign/malignant/unfavorable obstetric outcome) and currently under treatment at the U.O.C. of Gynecology and Pathophysiology of Human Reproduction Polyclinic S. Orsola-Malpighi and registered with the Italian Association for Androgen Insensitivity and Similar Conditions-AISIA.
* Informed consent
* Networked electronic device ensuring connection to the platform and subsequent questionnaire filling
* Internet network
* Personal email address, to which the link for filling out the questionnaires will be sent

Exclusion Criteria:

* no exclusion criteria are provided

Ages: 18 Years to 44 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The subjects to be enrolled in the study are patients taken care of at the U.O.C. of Gynecology and Pathophysiology of Human Reproduction Polyclinic S. Orsola-Malpighi and/or registered with the Italian Association for Androgen Insensitivity Syndrome and similar conditions-AISIA.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2021-04-05 (Actual); Primary Completion 2024-04-05 (Actual); Study Completion 2026-04-05 (Estimated)

PRIMARY OUTCOMES:
Questionnaire | 1 year
  In detail, the first part of the questionnaire contains a series of questions concerning socio-demographic aspects, pathological and family history, lifestyles, health status and perceived quality of life. In addition, the following structured and validated questionnaire will be required:
  - Brief Symptom Checklist-BSCL (Scale from 0 to 4)

CONTACTS AND LOCATIONS:
Overall Officials: Maria C Meriggiola, MD, Principal Investigator — IRCCS Bologna
Locations (1):
- IRCCS Azienda Ospedaliero-Unioversitaria di Bologna, Bologna, Bologna, Italy

IPD SHARING:
Plan to Share IPD: No